CLINICAL TRIAL: NCT05249127
Title: 64Cu-SAR-bisPSMA Positron Emission Tomography: A Phase 1/2 Study of Participants With Biochemical Recurrence of Prostate Cancer
Brief Title: 64Cu-SAR-bisPSMA for Identification of Participants With Recurrence of Prostate Cancer (COBRA)
Acronym: COBRA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clarity Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP06
Record Dates: First submitted 2022-02-02; First posted 2022-02-21 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-08

CONDITIONS: Biochemical Recurrence of Malignant Neoplasm of Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 64Cu-SAR-bisPSMA (Experimental): Patients will receive a single administration of 200 megabecquerels (MBq) of 64Cu-SAR-bisPSMA.
  Interventions: Drug: 64Cu-SAR-bisPSMA

INTERVENTIONS:
Drug: 64Cu-SAR-bisPSMA — 64Cu-SAR-bisPSMA

SUMMARY:
The aim of this study is to determine the safety and efficacy of 64Cu-SAR-bisPSMA and determine the ability of 64Cu-SAR-bisPSMA Positron emission tomography (PET)/computed tomography (CT) to correctly detect the recurrence of prostate cancer in participants with biochemical recurrence of prostate cancer following definitive therapy.

DETAILED DESCRIPTION:
Participants with biochemical evidence of recurrence of PC were evaluated with 64CU-SAR-bisPSMA PET/CT (Day 0 and Day 1) and by conventional methodologies up to 180 days later, eg. Histopathology/biopsy, conventional imaging, PSA reduction post focal salvage therapy or radiotherapy with no concomitant androgen deprivation therapy. Three independent central readers blinded to the participant number, the time of the PET/CT scan and the results of the conventional methodologies assessed the 64Cu-SAR-bisPSMA PET/CT. Three separate independent readers assessed the results of the conventional methodologies.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Signed informed consent.
3. Life expectancy ≥ 12 weeks as determined by the Investigator.
4. Histologically confirmed adenocarcinoma of prostate per original diagnosis and completed subsequent definitive therapy.
5. Suspected recurrence of prostate cancer (PC) based on rising Prostate-specific antigen (PSA) after definitive therapy on the basis of:

   1. Post-radical prostatectomy: Detectable or rising PSA that is ≥ 0.2 ng/mL with a confirmatory PSA ≥ 0.2 ng/mL (per American Urological Association recommendation) or
   2. Post-radiation therapy, cryotherapy, or brachytherapy: Increase in PSA level that is elevated by ≥ 2 ng/mL above the nadir (per American Society for Therapeutic Radiology and Oncology-Phoenix consensus definition).
6. Negative or equivocal findings for PC on conventional imaging performed as part of standard of care workup within 60 days prior to Day 0.
7. The Eastern Cooperative Oncology performance status 0-2.
8. Adequate recovery from acute toxic effects of any prior therapy.
9. Estimated Glomerular Filtration Rate of 30 mL/min or higher.
10. Adequate liver function.
11. For participants who have partners of childbearing potential: Partner and/or participant must use a method of birth control with adequate barrier protection.

Exclusion Criteria:

1. Participants who received other investigational agents within 28 days prior to Day 0.
2. Participants administered any high energy (>300 kiloelectronvolts (keV)) gamma-emitting radioisotope within 5 physical half-lives prior to Day 0.
3. Ongoing treatment or treatment within 90 days of Day 0 with any systemic therapy (e.g. androgen-deprivation therapy, antiandrogen, gonadotropin-releasing hormone, luteinizing hormone-releasing hormone agonist or antagonist) for PC.
4. Known or expected hypersensitivity to 64Cu-SAR-bisPSMA or any of its components.
5. Any serious medical condition or extenuating circumstance which the investigator feels may interfere with the procedures or evaluations of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Othon Gervasio, Study Director — Clarity Pharmaceuticals
Locations (5):
- United States (5):
  - Tower Urology, Los Angeles, California
  - GU Research Network, Omaha, Nebraska
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period:
  11 Apr 2022 to 23 Jan 2023
Groups:
- 64Cu-SAR-bisPSMA Injection: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR-bisPSMA followed by a PET/CT scan Day 0 (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Period: Overall Study
Arm/Group | 64Cu-SAR-bisPSMA Injection
Started | 52
Completed | 32
Not Completed | 20
Not completed — Protocol Violation | 13
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 2
Not completed — Participant Non-compliance | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received any amount of 64Cu-SAR-bisPSMA.
Arm/Group | 64Cu-SAR-bisPSMA Injection
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 49
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 52
Baseline PSA [Mean (Standard Deviation); unit: ng/mL] | 2.973 (4.1722)

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability
Description: Incidence and severity of Treatment-Emergent Adverse Events (TEAE) and Serious Adverse Events. Adverse Events were assessed by CTCAE version 5.0
Time Frame: up to 7 days post injection
Population: All Participants who received any amount of 64Cu-SAR-bisPSMA.
Measure: Count of Participants; unit: Participants
Arm/Group | 64Cu-SAR-bisPSMA Injection
Number analyzed (Participants) | 52
Participants
  Any TEAE | 10
  TEAE Grade 1 to 2 | 8
  TEAE Grade 3 | 2
  TEAE Grade 4 to 5 | 0
  TEAE Related to 64Cu-SAR-bisPSMA | 1
  Serious TEAE | 1
  Serious TEAE related to Cu64-SAR-bisPSMA | 0
  TEAE leading to withdrawal from study | 0
  TEAE with fatal outcome | 0

2. Primary Outcome: Participant-level Correct Detection Rate (CDR)- Day 0
Description: The percentage of TP participants on the Day 0 scan out of all participants with a Day 0 scan.
Time Frame: Day 0 (1- 4 hours) post injection
Population: All participants who received any amount of 64Cu-SAR-bisPSMA with 64Cu-SAR-bisPSMA PET/CT imaging results available from at least one central reader and had at least one evaluable reference datapoint (participant-level or region-level).
Measure: Number (95% Confidence Interval); unit: percentage of TP participants
Groups:
- 64Cu-SAR-bisPSMA: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR-bisPSMA followed by a PET/CT scan Day 0 (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | 64Cu-SAR-bisPSMA
Number analyzed (Participants) | 42
percentage of TP participants
  Reader 1 | 26.2 [13.9 to 42.0]
  Reader 2 | 23.8 [12.1 to 39.5]
  Reader 3 | 19.0 [8.6 to 34.1]

3. Primary Outcome: Participant-level CDR- Day 1
Description: The percentage of TP participants on the Day 1 scan out of all participants with a Day 1 scan.
Time Frame: Day 1 (24+/-6 Hours) post injection
Population: All participants who received any amount of 64Cu-SAR-bisPSMA with 64Cu-SAR-bisPSMA PET/CT imaging results available from at least one central reader and had at least one evaluable reference datapoint.
Measure: Number (95% Confidence Interval); unit: percentage of TP participants
Groups:
- 64Cu-SAR-bisPSMA PET Injection: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR-bisPSMA followed by a PET/CT scan Day 0 (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | 64Cu-SAR-bisPSMA PET Injection
Number analyzed (Participants) | 42
percentage of TP participants
  Reader 1 | 33.3 [19.6 to 49.5]
  Reader 2 | 33.3 [19.6 to 49.5]
  Reader 3 | 26.2 [13.9 to 42.0]

4. Primary Outcome: Region-level Positive Predictive Value (PPV)- Day 0
Description: The percentage of TP regions on the Day 0 scan out of all positive regions on the Day 0 scan.
Time Frame: Day 0 (1- 4 hours)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of TP regions
Units Other Than Participants: Regions
Arm/Group | 64Cu-SAR-bisPSMA Injection
Number analyzed (Participants) | 42
Number analyzed (Regions) | 195
percentage of TP regions
  Reader 1 | 41.2 [24.6 to 59.3]
  Reader 2 | 44.8 [26.4 to 64.3]
  Reader 3 | 39.1 [19.7 to 61.5]

5. Primary Outcome: Region-level PPV- Day 1
Description: The percentage of TP regions on the Day 1 scan out of all positive regions on the Day 1 scan.
Time Frame: Day 1 (24 +/- 6 hours)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of TP regions
Units Other Than Participants: Regions
Arm/Group | 64Cu-SAR-bisPSMA Injection
Number analyzed (Participants) | 42
Number analyzed (Regions) | 195
percentage of TP regions
  Reader 1 | 41.5 [26.3 to 57.9]
  Reader 2: number analyzed (Regions) | 194
  Reader 2 | 32.7 [20.3 to 47.1]
  Reader 3 | 43.3 [25.5 to 62.6]

6. Secondary Outcome: Biodistribution of 64Cu-SAR-bisPSMA- SUVmean
Description: The mean Standardized Uptake Value (SUVmean) in lesions, visceral soft tissue and bone.
Time Frame: Day 0 (1 -4 hours) and Day 1 (24 +/- 6 hours) post injection
Population: All enrolled participants who received any amount of 64Cu-SAR-bisPSMA who had at least one biodistribution measure. The number of participants analyzed varied depending on the number of lesions identified by each reader in each participant and in each region.
Measure: Mean (Standard Deviation); unit: g/mL
Groups:
- SUVmean- Day 0; SUVmean - Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | SUVmean- Day 0 | SUVmean - Day 1
Number analyzed (Participants) | 50 | 50
g/mL
  Reader 1 All Lesions: number analyzed (Participants) | 28 | 37
  Reader 1 All Lesions | 9.898 (5.9588) | 15.818 (15.0800)
  Reader 2 All Lesions: number analyzed (Participants) | 28 | 40
  Reader 2 All Lesions | 8.990 (5.8339) | 14.678 (19.4486)
  Reader 3 All Lesions: number analyzed (Participants) | 22 | 28
  Reader 3 All Lesions | 6.635 (3.2447) | 14.729 (11.1719)
  Reader 1 Bone Lesions: number analyzed (Participants) | 8 | 7
  Reader 1 Bone Lesions | 9.188 (4.7099) | 17.699 (10.7888)
  Reader 2 Bone Lesions: number analyzed (Participants) | 7 | 12
  Reader 2 Bone Lesions | 8.611 (4.2796) | 10.503 (11.9074)
  Reader 3 Bone Lesions: number analyzed (Participants) | 4 | 6
  Reader 3 Bone Lesions | 7.283 (4.4456) | 19.408 (10.9045)
  Reader 1 Soft Tissue Lesions: number analyzed (Participants) | 23 | 35
  Reader 1 Soft Tissue Lesions | 9.706 (6.2907) | 15.56 (15.5137)
  Reader 2 Soft Tissue Lesions: number analyzed (Participants) | 23 | 36
  Reader 2 Soft Tissue Lesions | 9.018 (6.1432) | 15.402 (20.2457)
  Reader 3 Soft Tissue Lesions: number analyzed (Participants) | 20 | 25
  Reader 3 Soft Tissue Lesions | 6.386 (3.2565) | 14.093 (11.4177)

7. Secondary Outcome: Biodistribution of 64Cu-SAR-bisPSMA- SUVmax
Description: SUVmax in lesions, visceral soft tissue and bone
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: g/mL
Groups:
- SUVmax- Day 0; SUVmax- Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | SUVmax- Day 0 | SUVmax- Day 1
Number analyzed (Participants) | 50 | 50
g/mL
  Reader 1 All Lesions: number analyzed (Participants) | 28 | 37
  Reader 1 All Lesions | 13.973 (8.9671) | 22.198 (18.6239)
  Reader 2 All Lesions: number analyzed (Participants) | 28 | 40
  Reader 2 All Lesions | 13.914 (10.3342) | 22.789 (32.3980)
  Reader 3 All Lesions: number analyzed (Participants) | 22 | 28
  Reader 3 All Lesions | 13.924 (7.6483) | 33.363 (37.7745)
  Reader 1 Bone Lesions: number analyzed (Participants) | 8 | 7
  Reader 1 Bone Lesions | 13.05 (6.4444) | 27.600 (17.7468)
  Reader 2 Bone Lesions: number analyzed (Participants) | 7 | 12
  Reader 2 Bone Lesions | 14.156 (6.0519) | 16.660 (17.9690)
  Reader 3 Bone Lesions: number analyzed (Participants) | 4 | 6
  Reader 3 Bone Lesions | 16.718 (5.0380) | 37.223 (19.9721)
  Reader 1 Soft Tissue Lesions: number analyzed (Participants) | 23 | 35
  Reader 1 Soft Tissue Lesions | 13.746 (9.5714) | 21.832 (19.2837)
  Reader 2 Soft Tissue Lesions: number analyzed (Participants) | 23 | 36
  Reader 2 Soft Tissue Lesions | 13.680 (11.1150) | 24.068 (33.7881)
  Reader 3 Soft Tissue Lesions: number analyzed (Participants) | 20 | 25
  Reader 3 Soft Tissue Lesions | 12.981 (8.1606) | 32.976 (39.5467)

8. Secondary Outcome: Biodistribution of 64Cu-SAR-bisPSMA- SUVr
Description: Lesion to Background ratio. SUVmax of the lesion divided by the SUVmean of gluteus background
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- SUVr - Day 0; SUVr - Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | SUVr - Day 0 | SUVr - Day 1
Number analyzed (Participants) | 50 | 50
ratio
  Reader 1 All Lesions: number analyzed (Participants) | 28 | 37
  Reader 1 All Lesions | 23.233 (14.0537) | 118.051 (90.7403)
  Reader 2 All Lesions: number analyzed (Participants) | 28 | 40
  Reader 2 All Lesions | 23.476 (17.3919) | 121.306 (160.9991)
  Reader 3 All Lesions: number analyzed (Participants) | 22 | 28
  Reader 3 All Lesions | 25.448 (15.0785) | 181.673 (171.6481)

9. Secondary Outcome: Participant-level PPV
Description: Percentage of TP participants on the Day 0 or Day 1 scan out of all participants with a positive Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of TP participants
Groups:
- Participant-level PPV- Day 0: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
- Participant-level PPV- Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer (PC) based on detectable or rising Prostate Specific Antigen (PSA) following definitive therapy, who had negative or equivocal findings on institutional standard of care (SOC) conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | Participant-level PPV- Day 0 | Participant-level PPV- Day 1
Number analyzed (Participants) | 42 | 42
percentage of TP participants
  Reader 1 | 44.0 [24.4 to 65.1] | 45.2 [27.3 to 64.0]
  Rader 2 | 43.5 [23.2 to 65.5] | 40.0 [23.9 to 57.9]
  Reader 3 | 42.1 [20.3 to 66.5] | 47.8 [26.8 to 69.4]

10. Secondary Outcome: Participant-level Detection Rate (DR)
Description: Percentage of participants with a positive Day 0 or Day 1 scan out of all participants with a Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours)
Population: All participants who received any amount of 64Cu-SAR-bisPSMA, and had 64Cu-SAR-bisPSMA PET/CT imaging results from at least one central reader
Measure: Number (95% Confidence Interval); unit: percentage of TP participants
Groups:
- Participant-level DR- Day 0; Participant-level DR- Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection)
Arm/Group | Participant-level DR- Day 0 | Participant-level DR- Day 1
Number analyzed (Participants) | 50 | 50
percentage of TP participants
  Reader 1 | 58.0 [43.2 to 71.8] | 74.0 [59.7 to 85.4]
  Reader 2 | 56.0 [41.3 to 70.0] | 80.0 [66.3 to 90.0]
  Reader 3 | 44.0 [30.0 to 58.7] | 58.0 [43.2 to 71.8]

11. Secondary Outcome: Participant-level False Positive Rate (FPR)
Description: Percentage of false positive (FP) participants on the Day 0 or Day 1 scan out of all participants with a positive Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of FP participants
Groups:
- Participant-level FPR- Day 0; Participant-level FPR- Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | Participant-level FPR- Day 0 | Participant-level FPR- Day 1
Number analyzed (Participants) | 42 | 42
percentage of FP participants
  Reader 1 | 53.8 [33.4 to 73.4] | 54.8 [36.0 to 72.7]
  Reader 2 | 54.2 [32.8 to 74.4] | 60.0 [42.1 to 76.1]
  Reader 3 | 57.9 [33.5 to 79.7] | 50.0 [29.1 to 70.9]

12. Secondary Outcome: Region-level FPR
Description: Percentage of FP regions on the Day 0 or Day 1 scan out of all positive regions on the Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/-6 hours)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of FP regions
Units Other Than Participants: regions
Groups:
- Region-level FPR-Day 0; Region-level FPR-Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | Region-level FPR-Day 0 | Region-level FPR-Day 1
Number analyzed (Participants) | 42 | 42
Number analyzed (regions) | 195 | 195
percentage of FP regions
  Reader 1 | 58.8 [40.7 to 75.4] | 57.1 [41.0 to 72.3]
  Reader 2: number analyzed (regions) | 195 | 194
  Reader 2 | 55.2 [35.7 to 73.6] | 67.3 [52.9 to 79.7]
  Reader 3 | 60.9 [38.5 to 80.3] | 56.7 [37.4 to 74.5]

13. Secondary Outcome: Participant-level Discrepant PET Negativity Rate
Description: Percentage of participants with contradicting Day 0 and Day 1 results for whom the Reference Standard was positive.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/-6 hours)
Population: All participants who received any amount of 64Cu-SAR-bisPSMA with 64Cu-SAR-bisPSMA PET/CT imaging results from at least one central reader and had a positive reference standard on the participant level.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 64Cu-SAR-bisPSMA Injection
Number analyzed (Participants) | 14
percentage of participants
  Reader 1 | 14.3 [1.8 to 42.8]
  Reader 2 | 21.4 [4.7 to 50.8]
  Reader 3 | 42.9 [17.7 to 71.1]

14. Secondary Outcome: Participant-level True Negative Rate (TNR)
Description: Percentage of TN participants on the Day 0 or Day 1 scan out of all participants with a negative Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/-6 hours)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of TN participants
Groups:
- Participant-level TNR- Day 0; Participant-level TNR- Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | Participant-level TNR- Day 0 | Participant-level TNR- Day 1
Number analyzed (Participants) | 42 | 42
percentage of TN participants
  Reader 1 | 50.0 [30.6 to 69.4] | 39.3 [21.5 to 59.4]
  Reader 2 | 53.6 [33.9 to 72.5] | 25.0 [10.7 to 44.9]
  Reader 3 | 60.7 [40.6 to 78.5] | 57.1 [37.2 to 91.8]

15. Secondary Outcome: Region-level TNR
Description: Percentage of TN regions on the Day 0 or Day 1 scan out of all negative regions on the Day 0 or Day 1 scan.
Time Frame: Day 0 (1-4 hours) and Day 1 (24 +/- 6 hours)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of TN regions
Units Other Than Participants: regions
Groups:
- Region-level TNR-Day 0; Region-level TNR- Day 1: Single Arm:
  Participants with suspected recurrence of prostate cancer based on detectable or rising PSA following definitive therapy, who had negative or equivocal findings on institutional standard of care conventional imaging, received a single intravenous Injection of 64Cu-SAR- bisPSMA followed by a PET/CT scan Day O (1 to 4 hours post injection) and Day 1 (24 +/- 6 hours post injection).
Arm/Group | Region-level TNR-Day 0 | Region-level TNR- Day 1
Number analyzed (Participants) | 42 | 42
Number analyzed (regions) | 195 | 195
percentage of TN regions
  Reader 1 | 88.7 [83.1 to 93.0] | 86.4 [80.5 to 91.1]
  Reader 2: number analyzed (regions) | 195 | 194
  Reader 2 | 91.0 [85.7 to 94.7] | 80.1 [73.4 to 85.7]
  Reader 3 | 92.1 [87.2 to 95.6] | 90.4 [85.1 to 94.3]

ADVERSE EVENTS:
Time Frame: Up to 7 days post injection
Description: Physical exam pre-dose and at Day 7. Vital signs pre and post dose and at Day 7. Duplicate 12-lead ECG pre and 30 +/- 10 minutes post dose. Hematology, biochemistry, urinalysis and coagulation lab tests at screening and 7 days post dose.
  Adverse event monitoring pre and post dose, and up to Day 7.
Groups:
- Safety Analysis Set: All participants enrolled who received any amount of 64Cu-SAR-bisPSMA.
Arm/Group | Safety Analysis Set
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52
Other Adverse Events (participants affected / at risk) | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set (N=52)
urosepsis (Infections and infestations) | 1 (1) — Grade 3 urosepsis. Serious criteria: hospitalization. Not related to 64Cu-SAR-bisPSMA. Commenced Day 3 post injection. Resolved in 5 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study results may only be published by the principal investigator / institution following the first multi-site publication. The proposed publication will be submitted to Sponsor at least 90 days prior to submission to the publication to allow the Sponsor to delete Sponsor Confidential Information (other than Study results), correct any inaccuracies or delay the publication to allow for filing of patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT05249127/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT05249127/SAP_002.pdf